CLINICAL TRIAL: NCT03395210
Title: An Adaptive, Open-Label, Dose-Finding, Phase 1/2 Study Investigating the Safety, Pharmacokinetics, and Clinical Activity of PRN1008, an Oral BTK Inhibitor, in Patients With Relapsed Immune Thrombocytopenia
Brief Title: A Study of Rilzabrutinib in Adult Patients With Immune Thrombocytopenia (ITP)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Principia Biopharma, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DFI17124; PRN1008-010 (Other: Principia Biopharma); U1111-1260-4044 (Registry Identifier: ICTRP); 2023-509397-39 (Registry Identifier: CTIS)
Record Dates: First submitted 2017-12-22; First posted 2018-01-10 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rilzabrutinib (PRN1008) Daily (Experimental): Part A approximately 60 patients: Up to 24 weeks open-label treatment with PRN1008 400mg BID; safety and dose evaluation. Patients who respond to PRN1008 per protocol may enter a long-term extension.
  Part B approximately 25 patients: Up to 24 weeks open-label treatment with PRN1008 400mg BID; safety and dose evaluation. Patients who respond to PRN1008 per protocol may enter a long-term extension
  Interventions: Drug: Rilzabrutinib

INTERVENTIONS:
Drug: Rilzabrutinib — BTK inhibitor
  Other Names: PRN1008

SUMMARY:
This was a 2 part (Part A and B) adaptive, open-label, dose-finding study of PRN1008 in patients with ITP who are refractory or relapsed with no available and approved therapeutic options, with a platelet count <30,000/μL on two counts no sooner than 7 days apart in the 15 days before treatment begins. The dose-finding portion of the study was completed. Part B treatment dose was 400 mg twice daily.

DETAILED DESCRIPTION:
This was a 2 part (Part A and B) adaptive, open-label, dose-finding study of PRN1008 in approximately 60 patients in Part A and approximately 25 patients in Part B.

Part A enrolled patients with ITP who were refractory or relapsed with no available and approved therapeutic options. Eligible patients had a platelet count <30,000/μL on two counts no sooner than 7 days apart in the 15 days before treatment begins. The active treatment period was 24 weeks and the post-treatment follow-up period is 4 weeks. In the dose-finding part of the study, each patient enrolled in the study was allowed to up-titrate their dose after 28 days of PRN1008 therapy, if they did not experience a platelet response or a dose-limiting toxicity (DLT) at the last dose level. Patients who responded to PRN1008 per protocol may enter a long term-extension.

Part B of the study included approximately 25 patients with ITP who had relapsed or had an insufficient response to prior therapies. Eligible patients had a platelet count <30,000/µL on two occasions no less than 7 days apart, within 15 days before treatment began and a platelet count of ≤35,000/µL on Study Day 1 (SD1). The study consisted of a 28-day screening period, 24-week active treatment period, and a long-term extension. After the last dose of PRN1008 there was a 4-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged 18 to 80 years old
* Immune-related ITP (both primary and secondary)

Exclusion Criteria:

* Pregnant or lactating women
* Current drug or alcohol abuse
* History of solid organ transplant
* Positive screening for HIV, hepatitis B, or hepatitis C

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2025-12-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Bandman, MD, Study Director — Principia Biopharma
Locations (31):
- United States (8):
  - Bleeding and Clotting Disorders Institute- Site Number : 1087, Peoria, Illinois
  - RCCA MC LLC- Site Number : 1091, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center- Site Number : 1092, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center- Site Number : 1099, Boston, Massachusetts
  - Mid Michigan Medical Center- Site Number : 1086, Midland, Michigan
  - New York Presbyterian Hospital/Weill Cornell Medical Center- Site Number : 1097, New York, New York
  - Pitt County Memorial Hospital- Site Number : 1095, Greenville, North Carolina
  - Seattle Cancer Care Alliance Site Number : 1098, Seattle, Washington
- Australia (6):
  - Investigational Site Number : 105, Canberra, Australian Capital Territory
  - Investigational Site Number : 104, Sydney, New South Wales
  - Investigational Site Number : 102, Woolloongabba, Queensland
  - Investigational Site Number : 101, Clayton, Victoria
  - Investigational Site Number : 106, Parkville, Victoria
  - Investigational Site Number : 103, Perth, Western Australia
- Bulgaria (3):
  - Investigational Site Number : 213, Pleven
  - Investigational Site Number : 214, Sofia
  - Investigational Site Number : 211, Varna
- Canada (2):
  - Investigational Site Number : 1161, Toronto, Ontario
  - Investigational Site Number : 1162, Montreal, Quebec
- Czechia (4):
  - Investigational Site Number : 431, Brno
  - Investigational Site Number : 433, Hradec Králové
  - Investigational Site Number : 434, Ostrava - Poruba
  - Investigational Site Number : 432, Prague
- Netherlands (2):
  - Investigational Site Number : 727, Rotterdam
  - Investigational Site Number : 728, The Hague
- Norway (2):
  - Investigational Site Number : 542, Bergen
  - Investigational Site Number : 541, Grålum
- United Kingdom (4):
  - Investigational Site Number : 981, Leicester, Leicestershire
  - Investigational Site Number : 983, London, London, City of
  - Investigational Site Number : 980, London, London, City of
  - Investigational Site Number : 984, Birmingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Cooper N, Jansen AJG, Bird R, Mayer J, Sholzberg M, Tarantino MD, Garg M, Ypma PF, McDonald V, Percy C, Kostal M, Goncalves I, Bogdanov LH, Gernsheimer TB, Diab R, Yao M, Daak A, Kuter DJ. Efficacy and Safety Results With Rilzabrutinib, an Oral Bruton Tyrosine Kinase Inhibitor, in Patients With Immune Thrombocytopenia: Phase 2 Part B Study. Am J Hematol. 2025 Mar;100(3):439-449. doi: 10.1002/ajh.27539. Epub 2025 Jan 22. PMID 39844469
- [Derived] Kuter DJ, Mayer J, Efraim M, Bogdanov LH, Baker R, Kaplan Z, Garg M, Trneny M, Choi PY, Jansen AJG, McDonald V, Bird R, Gumulec J, Kostal M, Gernsheimer T, Ghanima W, Daak A, Cooper N. Long-term treatment with rilzabrutinib in patients with immune thrombocytopenia. Blood Adv. 2024 Apr 9;8(7):1715-1724. doi: 10.1182/bloodadvances.2023012044. PMID 38386978
- [Derived] Kuter DJ, Efraim M, Mayer J, Trneny M, McDonald V, Bird R, Regenbogen T, Garg M, Kaplan Z, Tzvetkov N, Choi PY, Jansen AJG, Kostal M, Baker R, Gumulec J, Lee EJ, Cunningham I, Goncalves I, Warner M, Boccia R, Gernsheimer T, Ghanima W, Bandman O, Burns R, Neale A, Thomas D, Arora P, Zheng B, Cooper N. Rilzabrutinib, an Oral BTK Inhibitor, in Immune Thrombocytopenia. N Engl J Med. 2022 Apr 14;386(15):1421-1431. doi: 10.1056/NEJMoa2110297. PMID 35417637
- [Derived] Del Pozo Martin Y. 2021 ASH annual meeting. Lancet Haematol. 2022 Feb;9(2):e92-e93. doi: 10.1016/S2352-3026(21)00384-7. Epub 2021 Dec 16. No abstract available. PMID 34922648
- See also: DFI17124 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26252&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 31 active centers in 8 countries. As prespecified in statistical analysis plan (SAP), Part A results were presented by either of the of the treatment group labels: Starting dose level (each participant was assigned to only one of the groups), dose level (dose received during the defined period. As most patients received more than one dose, a given patient could be assigned to multiple dose levels) and overall.
Pre-assignment Details: A total of 60 participants in Part A and 26 participants in Part B were enrolled in the study. The results are presented up to primary completion date 31 January 2023.
Groups:
- Part A: Starting Dose 200 mg QD: Participants received rilzabrutinib 200 milligrams (mg) orally once daily (QD) as starting dose from Day 1 to 4 weeks. Participants were allowed to up-titrate the dose levels unless withdrawn, had a platelet response to current dose level, or the next dose level had been determined to be ineligible for further enrollment every 4 weeks up to the maximum allowed 400 mg twice daily (BID) (800 mg/day) over 24 weeks of treatment period.
- Part A: Starting Dose 400 mg QD: Participants received rilzabrutinib 400 mg orally QD as starting dose from Day 1 to 4 weeks. Participants were allowed to up-titrate the dose levels unless withdrawn, had a platelet response to current dose level, or the next dose level had been determined to be ineligible for further enrollment every 4 weeks up to the maximum allowed 400 mg BID (800 mg/day) over 24 weeks of treatment period.
- Part A: Starting Dose 300 mg BID: Participants received rilzabrutinib 300 mg orally BID as starting dose from Day 1 to 4 weeks. Participants were allowed to up-titrate the dose levels unless withdrawn, had a platelet response to current dose level, or the next dose level had been determined to be ineligible for further enrollment every 4 weeks up to the maximum allowed 400 mg BID (800 mg/day) over 24 weeks of treatment period.
- Part A: Starting Dose 400 mg BID: Participants received rilzabrutinib 400 mg orally BID as starting dose from Day 1 to 24 weeks, unless withdrawn or had a platelet response to current dose level.
- Part B: Rilzabrutinib 400 mg BID: Participants received rilzabrutinib 400 mg orally BID from Day 1 up to 24 weeks of treatment period.
Period: Overall Study
Arm/Group | Part A: Starting Dose 200 mg QD | Part A: Starting Dose 400 mg QD | Part A: Starting Dose 300 mg BID | Part A: Starting Dose 400 mg BID | Part B: Rilzabrutinib 400 mg BID
Started | 9 | 1 | 5 | 45 | 26
Completed | 4 | 0 | 0 | 15 | 4
Not Completed | 5 | 1 | 5 | 30 | 22
Not completed — Other | 0 | 0 | 0 | 0 | 1
Not completed — Participant Uncooperative or Noncompliant | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 2 | 4 | 3
Not completed — Need of Rescue Medication | 1 | 0 | 1 | 4 | 0
Not completed — Lack of Response | 0 | 0 | 0 | 5 | 5
Not completed — Participant was Erroneously Enrolled in the Study | 1 | 0 | 0 | 0 | 1
Not completed — Participant Decision | 1 | 1 | 0 | 4 | 0
Not completed — Ongoing at the Time of Primary Completion Date | 1 | 0 | 2 | 13 | 11

BASELINE CHARACTERISTICS:
Population: Part A: Intent-to-treat population (ITT) consisted of all participants who had enrolled into the study.
  Part B: The enrolled population consisted of all participants from screened population (who signed informed consent) who had been allocated to rilzabrutinib regardless of whether rilzabrutinib was received or not.
Groups:
- Part A: Starting Dose 200 mg QD: Participants received rilzabrutinib 200 mg orally QD as starting dose from Day 1 to 4 weeks. Participants were allowed to up-titrate the dose levels unless withdrawn, had a platelet response to current dose level, or the next dose level had been determined to be ineligible for further enrollment every 4 weeks up to the maximum allowed 400 mg BID (800 mg/day) over 24 weeks of treatment period.
- Total: Total of all reporting groups
Arm/Group | Part A: Starting Dose 200 mg QD | Part A: Starting Dose 400 mg QD | Part A: Starting Dose 300 mg BID | Part A: Starting Dose 400 mg BID | Part B: Rilzabrutinib 400 mg BID | Total
Number analyzed (Participants) | 9 | 1 | 5 | 45 | 26 | 86
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 8 | 1 | 5 | 38 | 19 | 71
  >= 65 years | 1 | 0 | 0 | 7 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 3 | 27 | 16 | 50
  Male | 5 | 1 | 2 | 18 | 10 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 1 | 5 | 39 | 21 | 75
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percentage of Participants Who Achieved 2 or More Consecutive Platelet Counts by Starting Dose Level and Overall
Description: The percentage of participants who achieved 2 or more consecutive platelet counts, separated by at least 5 days, of >=50,000/ microliter (μL) and an increase of platelet count of >=20,000/μL from baseline, by starting dose level and overall, without use of rescue medication in the 4 weeks prior to the latest elevated platelet count. 95% confidence interval (CI) was based on the Clopper-Pearson method. The average of the 2 screening results and the Cycle 1 Day 1 result were used as the baseline value.
Time Frame: Up to 24 Weeks
Population: ITT population consisted of all participants who had enrolled into the study. It was prespecified (SAP), data was analyzed by overall and starting dose level.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part A: Overall: All participants who received rilzabrutinib (200 mg QD or 400 mg QD or 300 mg BID or 400 mg BID) at all dose levels over 24 weeks of treatment period, unless withdrawn or had a platelet response to dose level.
Arm/Group | Part A: Starting Dose 200 mg QD | Part A: Starting Dose 400 mg QD | Part A: Starting Dose 300 mg BID | Part A: Starting Dose 400 mg BID | Part A: Overall
Number analyzed (Participants) | 9 | 1 | 5 | 45 | 60
percentage of participants | 44.4 [13.70 to 78.80] | 0.0 [0.00 to 97.50] | 40.0 [5.27 to 85.34] | 40.0 [25.70 to 55.67] | 40.0 [27.56 to 53.46]

2. Primary Outcome: Part B: Percentage of Participants Who Achieved Platelet Counts >=50,000/μL
Description: The percentage of participants who achieved platelet counts >=50,000/μL on at least 8 out of the last 12 weeks of the 24-week treatment period without the use of rescue medication after 10 weeks of active treatment. 95% CI was based on the Clopper-Pearson exact method.
Time Frame: Up to 24 Weeks
Population: ITT population consisted of all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: Rilzabrutinib 400 mg BID
Number analyzed (Participants) | 26
percentage of participants | 34.6 [17.21 to 55.67]

3. Primary Outcome: Part A: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment Related Treatment-Emergent Adverse Events
Description: Adverse event (AE): any untoward medical occurrence in participant or clinical study participant, temporally associated with the use of rilzabrutinib, whether or not considered related to rilzabrutinib. TEAEs: AEs that developed or worsened or became serious on or after the first dose administration of rilzabrutinib (Day 1). Any TEAEs are considered treatment-related TEAEs as per Investigator's evaluation of participant's circumstances surrounding the event, and an evaluation of any potential alternative causes to determine whether an TEAE can be considered as related to the rilzabrutinib.
Time Frame: From first dose of rilzabrutinib (Day 1) up to last dose + 1 (up to 294 days)
Population: Safety population consisted of all participants who received at least 1 dose of rilzabrutinib. It was prespecified (SAP), data was analyzed by overall and dose level and participants could be classified into multiple dose levels.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Dose Level 200 mg QD: All participants who received rilzabrutinib 200 mg orally QD over 24 weeks of treatment period, unless withdrawn or had a platelet response to current dose level.
- Part A: Dose Level 400 mg QD: All participants who received rilzabrutinib 400 mg orally QD over 24 weeks of treatment period, unless withdrawn or had a platelet response to current dose level.
- Part A: Dose Level 300 mg BID: All participants who received rilzabrutinib 300 mg orally BID over 24 weeks of treatment period, unless withdrawn or had a platelet response to current dose level.
- Part A: Dose Level 400 mg BID: All participants who received rilzabrutinib 400 mg orally BID over 24 weeks of treatment period, unless withdrawn or had a platelet response to current dose level.
Arm/Group | Part A: Dose Level 200 mg QD | Part A: Dose Level 400 mg QD | Part A: Dose Level 300 mg BID | Part A: Dose Level 400 mg BID | Part A: Overall
Number analyzed (Participants) | 9 | 8 | 12 | 52 | 60
Participants
  TEAEs | 3 | 3 | 5 | 44 | 48
  Treatment related TEAEs | 2 | 2 | 2 | 29 | 31

4. Primary Outcome: Part B: Number of Participants With Treatment-Emergent Adverse Events and Treatment Related Treatment-Emergent Adverse Events
Description: AE any untoward medical occurrence in participant or clinical study participant, temporally associated with the use of rilzabrutinib, whether or not considered related to rilzabrutinib. TEAEs: AEs that developed or worsened or became serious during the treatment-emergent period, defined as any time after the first dose administration of rilzabrutinib (Day 1). Any TEAEs are considered treatment-related TEAEs as per Investigator's evaluation of participant's circumstances surrounding the event, and an evaluation of any potential alternative causes to determine whether an TEAE can be considered as related to rilzabrutinib.
Time Frame: From first dose of rilzabrutinib (Day 1) up to last dose + 1 (approximately 170 days)
Population: Safety population consisted of all participants who had taken rilzabrutinib, regardless of the amount administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Rilzabrutinib 400 mg BID
Number analyzed (Participants) | 26
Participants
  TEAEs | 22
  Treatment related TEAEs | 16

5. Secondary Outcome: Part A: Percentage of Weeks With Platelet Counts >=50,000/μL by Starting Dose Level and Overall
Description: The percentage of weeks in which participants achieved platelet counts >=50,000/μL in the treatment period are summarized here.
Time Frame: Up to 24 Weeks
Population: ITT population consisted of all participants who had enrolled into the study. Only participants with data collected at specified timepoints are reported. It was prespecified (SAP), data was analyzed by overall and starting dose level.
Measure: Mean (Standard Deviation); unit: percentage of weeks
Arm/Group | Part A: Starting Dose 200 mg QD | Part A: Starting Dose 400 mg QD | Part A: Starting Dose 300 mg BID | Part A: Starting Dose 400 mg BID | Part A: Overall
Number analyzed (Participants) | 8 | 1 | 5 | 45 | 59
percentage of weeks | 27.92 (29.42) | 0.00 (NA) — Standard deviation (SD) cannot be calculated for a single participant. | 39.58 (41.30) | 28.14 (36.41) | 28.60 (35.39)

6. Secondary Outcome: Part A: Percentage of Participants With 4 Out of the Final 8 Platelet Counts >=50,000/μL by Starting Dose Level and Overall
Description: The percentage of participants who had at least 4 out of the final 8 platelet counts >=50,000/μL are summarized here. The final 8 scheduled platelet counts are the measurements performed in the last 8 weeks of rilzabrutinib (depending on treatment duration, not necessarily from Week 19 to Week 24) in the treatment period. 95% CI was based on the Clopper-Pearson method.
Time Frame: Up to 24 Weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Starting Dose 200 mg QD | Part A: Starting Dose 400 mg QD | Part A: Starting Dose 300 mg BID | Part A: Starting Dose 400 mg BID | Part A: Overall
Number analyzed (Participants) | 9 | 1 | 5 | 45 | 60
percentage of participants | 11.1 [0.28 to 48.25] | 0.0 [0.00 to 97.50] | 40.0 [5.27 to 85.34] | 31.1 [18.17 to 46.65] | 28.3 [17.45 to 41.44]

7. Secondary Outcome: Part A: Change From Baseline to the Average of Post Day 1 Platelet Counts by Dose Level and Overall
Description: Average of post Day 1 platelet count is equivalent to average of (average of each participant's post-Day 1 platelet counts), included platelet counts up to 1 day after the date of last dose of rilzabrutinib and excluded platelet counts on or after date of rescue, if applicable. The average of the 2 screening results and the Cycle 1 Day 1 result measured on different date were used as the baseline value.
Time Frame: Baseline and up to 24 Weeks
Population: ITT population consisted of all participants who had enrolled into the study. It was prespecified (SAP), data was analyzed by overall and dose level and participants can be classified into multiple dose levels. Only participants with data who had more than 4 weeks of rilzabrutinib within a dose level are reported in each dose level. Participants with more than 4 weeks of study drug across all dose levels are included in overall.
Measure: Mean (Standard Deviation); unit: platelets x10^9/Liter (L)
Arm/Group | Part A: Dose Level 200 mg QD | Part A: Dose Level 400 mg QD | Part A: Dose Level 300 mg BID | Part A: Dose Level 400 mg BID | Part A: Overall
Number analyzed (Participants) | 3 | 1 | 6 | 45 | 54
platelets x10^9/Liter (L) | 6.92 (22.52) | 68.10 (NA) — SD cannot be calculated for a single participant. | 37.05 (29.10) | 29.92 (41.70) | 28.61 (39.57)

8. Secondary Outcome: Part A: Number of Weeks With Platelet Counts >=50,000/μL by Starting Dose Level and Overall
Description: The number of weeks in which participant achieved platelet counts >=50,000/μL in the treatment period are summarized here. The number of weeks is based on the number of scheduled weekly assessments, by study day.
Time Frame: Up to 24 Weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Part A: Starting Dose 200 mg QD | Part A: Starting Dose 400 mg QD | Part A: Starting Dose 300 mg BID | Part A: Starting Dose 400 mg BID | Part A: Overall
Number analyzed (Participants) | 8 | 1 | 5 | 45 | 59
weeks | 5.9 (7.8) | 0.0 (NA) — SD cannot be calculated for a single participant. | 10.2 (12.0) | 5.7 (8.1) | 6.0 (8.3)

9. Secondary Outcome: Part A: Number of Weeks With Platelet Counts >=30,000/μL by Starting Dose Level and Overall
Description: The number of weeks in which participant achieved platelet counts >=30,000/μL in the treatment period are summarized here. The number of weeks is based on the number of scheduled weekly assessments, by study day.
Time Frame: Up to 24 Weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Part A: Starting Dose 200 mg QD | Part A: Starting Dose 400 mg QD | Part A: Starting Dose 300 mg BID | Part A: Starting Dose 400 mg BID | Part A: Overall
Number analyzed (Participants) | 8 | 1 | 5 | 45 | 59
weeks | 8.4 (11.2) | 0.0 (NA) — SD cannot be calculated for a single participant. | 14.0 (14.1) | 8.8 (9.2) | 9.0 (9.8)

10. Secondary Outcome: Part A: Time to First Platelet Count >=50,000/μL Across All Dose Levels
Description: Time to first platelet count >=50,000/μL during the treatment period in days was calculated as: (date of first occurrence of platelet count >=50,000/μL - date of first rilzabrutinib dosing) +1.
Time Frame: Up to 24 Weeks
Population: ITT population consisted of all participants who had enrolled into the study. It was prespecified (protocol and SAP) that data will be analyzed for overall across all dose levels, so combined data reported here. Only participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Part A: Overall Participants: All participants who received rilzabrutinib (200 mg QD or 400 mg QD or 300 mg BID or 400 mg BID) at all dose levels over 24 weeks of treatment period, unless withdrawn or had a platelet response to dose level.
Arm/Group | Part A: Overall Participants
Number analyzed (Participants) | 30
days | 27.4 (31.86)

11. Secondary Outcome: Part B: Number of Weeks With Platelet Counts >= 50,000/μL or >= 30,000/μL and Doubling the Baseline
Description: The number of weeks in which participant achieved platelet counts with thresholds as: >=50,000/μL or >=30,000/μL and doubling the baseline in the absence of rescue therapy (platelet counts will be censored for 4 weeks after the use of rescue medication, if given) are summarized here. Baseline is defined as the average of 3 platelet counts: 2 qualified screening platelet counts collected in electronic case report form (eCRF) and Week 1 (study day 1) platelet count.
Time Frame: Up to 24 Weeks
Population: ITT population consisted of all enrolled participants.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Part B: Rilzabrutinib 400 mg BID
Number analyzed (Participants) | 26
weeks | 9.3 (10.1)

12. Secondary Outcome: Part B: Percentage of Participants Who Achieved 2 or More Consecutive Platelet Counts
Description: Percentage of participants who achieved 2 or more consecutive platelet counts, separated by at least 5 days, of >=50,000/μL and an increase of platelet count of >=20,000/μL from baseline without use of rescue medication in the 4 weeks prior to the latest elevated platelet count are summarized here. Baseline is defined as the average of 3 platelet counts: 2 qualified screening platelet counts collected in eCRF and Week 1 (study day 1) platelet count. 95% CI was based on the Clopper-Pearson exact method.
Time Frame: Up to 24 Weeks
Population: ITT population consisted of all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: Rilzabrutinib 400 mg BID
Number analyzed (Participants) | 26
percentage of participants | 42.3 [23.35 to 63.08]

13. Secondary Outcome: Part B: Number of Weeks With Platelet Counts >=30,000/μL and Doubling the Baseline
Description: The number of weeks in which participant achieved platelet counts >=30,000/μL and doubling the baseline in the absence of rescue therapy (platelet counts will be censored for 4 weeks after the use of rescue medication, if given) are summarized here. Baseline is defined as the average of 3 platelet counts: 2 qualified screening platelet counts collected in eCRF and Week 1 (study day 1) platelet count.
Time Frame: Up to 24 Weeks
Population: ITT population consisted of all enrolled participants.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Part B: Rilzabrutinib 400 mg BID
Number analyzed (Participants) | 26
weeks | 9.3 (10.1)

14. Secondary Outcome: Part B: Percentage of Participants Who Received Rescue Medication
Description: Rescue medication is defined as any therapy used to rescue a participant (1 of intravenous immunoglobulin [IVIG], high-dose steroids, platelet infusion or anti-D immunoglobulin infusion). Percentage of participants who received rescue medication are summarized here. 95% CI was based on the Clopper-Pearson exact method.
Time Frame: Up to 24 Weeks
Population: ITT population consisted of all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: Rilzabrutinib 400 mg BID
Number analyzed (Participants) | 26
percentage of participants | 11.5 [2.45 to 30.15]

15. Secondary Outcome: Part B: Change From Baseline in Idiopathic Thrombocytopenic Purpura Bleeding Scale (IBLS)
Description: The IBLS is a bleeding assessment score. IBLS comprises of 11 sites for female and 10 sites for male, and each site is scored from 0 (none) to 2 (marked bleeding). The total overall score ranges from 0-22, with higher scores indicating higher presence of marked bleeding. For each participant, an IBLS score at each visit was calculated by taking the average across 11 items (10 for male and postmenopausal women) at 9 anatomical sites (8 for male and postmenopausal women). For each participant, a mean IBLS score was also calculated by taking the average across all post-baseline visits during the 24-week treatment period. IBLS average value ranges from 0 to 2. The smaller the IBLS average value is, the healthier the participants are. For change from baseline, negative value indicates an improvement. The baseline value is defined as the last available value before the first dose rilzabrutinib.
Time Frame: Baseline and up to 24 weeks
Population: ITT population consisted of all enrolled participants. Only participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Rilzabrutinib 400 mg BID
Number analyzed (Participants) | 24
score on a scale | -0.07 (0.13)

16. Secondary Outcome: Part A: Percentage of Participants Who Received Rescue Medication by Dose Levels and Overall
Description: Rescue medication is defined as any therapy used to rescue a participant (1 of IVIG, high-dose steroids, platelet infusion or anti-D immunoglobulin infusion). The percentage of participants who received rescue medication for each dose level and overall are summarized here. 95% CI was based on the Clopper-Pearson method.
Time Frame: Up to 24 Weeks
Population: Safety population consisted of all participants who received at least 1 dose of rilzabrutinib. Participants are classified into different dose levels according to the dose received at the start of rescue medication. A given participant can be classified into multiple dose levels. It was prespecified (SAP), data was analyzed by overall and dose level.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Dose Level 200 mg QD | Part A: Dose Level 400 mg QD | Part A: Dose Level 300 mg BID | Part A: Dose Level 400 mg BID | Part A: Overall
Number analyzed (Participants) | 9 | 8 | 12 | 52 | 60
percentage of participants | 11.1 [0.28 to 48.25] | 0.0 [0.00 to 36.94] | 8.3 [0.21 to 38.48] | 9.6 [3.20 to 21.03] | 11.7 [4.82 to 22.57]

17. Secondary Outcome: Part A: Percentage of Participants With Grade 2 or Higher Bleeding Event by Dose Level and Overall
Description: The percentage of participants with intensity grade 2 or higher bleeding event are summarized for each dose level and overall. The TEAEs with standardized medical dictionary for regulatory activities (MedDRA) query (SMQ) hemorrhages were medically determined for analysis of bleeding events. 95% CI was based on the Clopper-Pearson method.
Time Frame: Up to 24 Weeks
Population: Safety population consisted of all participants who received at least 1 dose of rilzabrutinib. Participants are classified into different dose levels according to the dose received at the start of the bleeding event. A given participant can be classified into multiple dose levels. It was prespecified (SAP), data was analyzed by overall and dose level.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Dose Level 200 mg QD | Part A: Dose Level 400 mg QD | Part A: Dose Level 300 mg BID | Part A: Dose Level 400 mg BID | Part A: Overall
Number analyzed (Participants) | 9 | 8 | 12 | 52 | 60
percentage of participants | 0.0 [0.00 to 33.63] | 0.0 [0.00 to 36.94] | 8.3 [0.21 to 38.48] | 17.3 [8.23 to 30.33] | 16.7 [8.29 to 28.52]

18. Secondary Outcome: Part A: Number of Participants With Idiopathic Thrombocytopenic Purpura/Immune Thrombocytopenia (ITP) Bleeding Assessment Tool (ITP-BAT) Scale by Dose Level
Description: The ITP-BAT scale comprises of 11 grades from 0 (none) to 2 (marked bleeding), with higher scores indicating higher presence of marked bleeding, assessed at 9 anatomical sites (skin, oral, epistaxis, gastrointestinal [GI], urinary, gynecological [GYN], pulmonary, intracranial hemorrhage [HEM], subconjunctival HEM) by history over the previous week (Hx). In addition, 2 sites (skin and oral), were also assessed by physical examination (PE). The 'worst ever' bleeding experienced at each site was graded using the same system. Here, 0 indicates none; 1 indicates 1-5 bruises and/or scattered petechiae and 2 indicates >5 bruises with size >2 centimeter (cm) and/or diffuse petechiae. Each participant summed up the transformed scores across all 11 sites per visit assessment. The total overall score ranges from 0-22 with the higher score indicating worst outcome.
Time Frame: Up to 24 Weeks
Population: Safety population consisted of all participants who received at least 1 dose of rilzabrutinib. It was prespecified (SAP), data was analyzed by dose level and participants can be classified into multiple dose levels.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Dose Level 200 mg QD | Part A: Dose Level 400 mg QD | Part A: Dose Level 300 mg BID | Part A: Dose Level 400 mg BID
Number analyzed (Participants) | 9 | 8 | 12 | 52
Participants
  Skin (PE): Score 0 | 7 | 8 | 6 | 32
  Skin (PE): Score 1 | 0 | 0 | 3 | 12
  Skin (PE): Score 2 | 0 | 0 | 0 | 6
  Skin (PE): Scoring not done/missing | 2 | 0 | 3 | 2
  Oral (PE): Score 0 | 7 | 8 | 9 | 42
  Oral (PE): Score 1 | 0 | 0 | 0 | 4
  Oral (PE): Score 2 | 0 | 0 | 0 | 4
  Oral (PE): Scoring not done/missing | 2 | 0 | 3 | 2
  Skin (Hx): Score 0 | 7 | 8 | 5 | 34
  Skin (Hx): Score 1 | 0 | 0 | 4 | 11
  Skin (Hx): Score 2 | 0 | 0 | 0 | 5
  Skin (Hx): Scoring not done/missing | 2 | 0 | 3 | 2
  Oral (Hx): Score 0 | 7 | 8 | 9 | 43
  Oral (Hx): Score 1 | 0 | 0 | 0 | 2
  Oral (Hx): Score 2 | 0 | 0 | 0 | 5
  Oral (Hx): Scoring not done/missing | 2 | 0 | 3 | 2
  Epistaxis: Score 0 | 7 | 8 | 9 | 49
  Epistaxis: Score 1 | 0 | 0 | 0 | 0
  Epistaxis: Score 2 | 0 | 0 | 0 | 1
  Epistaxis: Scoring not done/missing | 2 | 0 | 3 | 2
  GI: Score 0 | 7 | 8 | 10 | 49
  GI: Score 1 | 0 | 0 | 0 | 1
  GI: Score 2 | 0 | 0 | 0 | 0
  GI: Scoring not done/missing | 2 | 0 | 2 | 2
  Urinary: Score 0 | 7 | 8 | 9 | 48
  Urinary: Score 1 | 0 | 0 | 0 | 2
  Urinary: Score 2 | 0 | 0 | 0 | 0
  Urinary: Scoring not done/missing | 2 | 0 | 3 | 2
  GYN: Score 0 | 1 | 1 | 4 | 22
  GYN: Score 1 | 0 | 0 | 0 | 1
  GYN: Score 2 | 0 | 0 | 0 | 1
  GYN: Scoring not done/missing | 8 | 7 | 8 | 28
  Pulmonary: Score 0 | 6 | 8 | 8 | 49
  Pulmonary: Score 1 | 0 | 0 | 0 | 0
  Pulmonary: Score 2 | 0 | 0 | 0 | 0
  Pulmonary: Scoring not done/missing | 3 | 0 | 4 | 3
  Intracranial HEM: Score 0 | 7 | 8 | 8 | 49
  Intracranial HEM: Score 1 | 0 | 0 | 0 | 0
  Intracranial HEM: Score 2 | 0 | 0 | 0 | 0
  Intracranial HEM: Scoring not done/missing | 2 | 0 | 4 | 3
  Subconjunctival HEM: Score 0 | 7 | 8 | 8 | 50
  Subconjunctival HEM: Score 1 | 0 | 0 | 0 | 0
  Subconjunctival HEM: Score 2 | 0 | 0 | 0 | 0
  Subconjunctival HEM: Scoring not done/missing | 2 | 0 | 4 | 2

19. Secondary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) of Rilzabrutinib
Description: Plasma samples were collected at specified timepoints to determine Cmax of rilzabrutinib.
Time Frame: Day 1 of Cycles 1, 2, 3, and 5 (each cycle 28 days)
Population: ITT population consisted of all participants who had enrolled into the study. It was prespecified (SAP), data was analyzed based on frequent sampling on Day 1 of a new, higher dosing level and reported by dose. Only participants who received rilzabrutinib with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A: Dose Level 200 mg QD | Part A: Dose Level 400 mg QD | Part A: Dose Level 300 mg BID | Part A: Dose Level 400 mg BID
Number analyzed (Participants) | 9 | 7 | 9 | 43
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 9 | 0 | 5 | 43
  Cycle 1 Day 1 | 154 (117) |  | 287 (149) | 273 (203)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 7 | 0 | 3
  Cycle 2 Day 1 |  | 451 (408) |  | 396 (257)
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 9 | 0
  Cycle 3 Day 1 |  |  | 319 (266) |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 2
  Cycle 5 Day 1 |  |  |  | 447 (67.2)

20. Secondary Outcome: Part A: Time of Observed Maximum Plasma Concentration (Tmax) of Rilzabrutinib
Description: Plasma samples were collected at specified timepoints to determine tmax of rilzabrutinib.
Time Frame: Day 1 of Cycles 1, 2, 3, and 5 (each cycle 28 days)
Population: as for outcome 19
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Part A: Dose Level 200 mg QD | Part A: Dose Level 400 mg QD | Part A: Dose Level 300 mg BID | Part A: Dose Level 400 mg BID
Number analyzed (Participants) | 9 | 7 | 9 | 43
hours (h)
  Cycle 1 Day 1: number analyzed (Participants) | 9 | 0 | 5 | 43
  Cycle 1 Day 1 | 1.43 [0.500 to 2.00] |  | 1.50 [1.00 to 1.53] | 1.50 [0.500 to 4.00]
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 7 | 0 | 3
  Cycle 2 Day 1 |  | 2.00 [1.00 to 3.03] |  | 1.05 [0.500 to 2.00]
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 9 | 0
  Cycle 3 Day 1 |  |  | 1.50 [0.500 to 3.00] |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 2
  Cycle 5 Day 1 |  |  |  | 1.25 [1.00 to 1.50]

21. Secondary Outcome: Part A: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Rilzabrutinib
Description: Plasma samples were collected at specified timepoints to determine AUClast of rilzabrutinib.
Time Frame: Day 1 of Cycles 1, 2, 3, and 5 (each cycle 28 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part A: Dose Level 200 mg QD | Part A: Dose Level 400 mg QD | Part A: Dose Level 300 mg BID | Part A: Dose Level 400 mg BID
Number analyzed (Participants) | 9 | 7 | 9 | 43
h*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 9 | 0 | 5 | 43
  Cycle 1 Day 1 | 320 (217) |  | 616 (334) | 642 (435)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 7 | 0 | 3
  Cycle 2 Day 1 |  | 986 (646) |  | 1150 (1030)
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 9 | 0
  Cycle 3 Day 1 |  |  | 788 (610) |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 2
  Cycle 5 Day 1 |  |  |  | 872 (412)

22. Secondary Outcome: Part A: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUCinf) of Rilzabrutinib
Description: Plasma samples were collected at specified timepoints to determine AUCinf of rilzabrutinib.
Time Frame: Day 1 of Cycles 1, 2, and 3 (each cycle 28 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part A: Dose Level 200 mg QD | Part A: Dose Level 400 mg QD | Part A: Dose Level 300 mg BID | Part A: Dose Level 400 mg BID
Number analyzed (Participants) | 9 | 5 | 7 | 35
h*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 9 | 0 | 5 | 35
  Cycle 1 Day 1 | 331 (224) |  | 653 (351) | 703 (455)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 5 | 0 | 1
  Cycle 2 Day 1 |  | 787 (446) |  | 827 (NA) — SD cannot be calculated for a single participant.
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 7 | 0
  Cycle 3 Day 1 |  |  | 818 (671) |

23. Secondary Outcome: Part A: Elimination Half-Life (t1/2) of Rilzabrutinib
Description: Plasma samples were collected at specified timepoints to determine t1/2 of rilzabrutinib.
Time Frame: Day 1 of Cycles 1, 2, and 3 (each cycle 28 days)
Population: as for outcome 19
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: Dose Level 200 mg QD | Part A: Dose Level 400 mg QD | Part A: Dose Level 300 mg BID | Part A: Dose Level 400 mg BID
Number analyzed (Participants) | 9 | 6 | 7 | 37
hours
  Cycle 1 Day 1: number analyzed (Participants) | 9 | 0 | 5 | 37
  Cycle 1 Day 1 | 1.36 [1.09 to 1.50] |  | 1.30 [1.15 to 1.95] | 1.32 [0.780 to 3.24]
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 6 | 0 | 1
  Cycle 2 Day 1 |  | 1.52 [1.17 to 3.89] |  | 1.34 [1.34 to 1.34]
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 7 | 0
  Cycle 3 Day 1 |  |  | 1.60 [1.18 to 1.88] |

24. Secondary Outcome: Part A: Apparent Volume of Distribution of the Drug After Oral Administration (Vz/F) of Rilzabrutinib
Description: Plasma samples were collected at specified timepoints to determine Vz/F of rilzabrutinib.
Time Frame: Day 1 of Cycles 1, 2, and 3 (each cycle 28 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Part A: Dose Level 200 mg QD | Part A: Dose Level 400 mg QD | Part A: Dose Level 300 mg BID | Part A: Dose Level 400 mg BID
Number analyzed (Participants) | 9 | 5 | 7 | 35
Liters
  Cycle 1 Day 1: number analyzed (Participants) | 9 | 0 | 5 | 35
  Cycle 1 Day 1 | 1780 (1180) |  | 1180 (611) | 1720 (1460)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 5 | 0 | 1
  Cycle 2 Day 1 |  | 2090 (2640) |  | 934 (NA) — SD cannot be calculated for a single participant.
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 7 | 0
  Cycle 3 Day 1 |  |  | 1650 (1510) |

25. Secondary Outcome: Part A: Apparent Total Clearance of the Drug From Plasma After Oral Administration (CL/F) of Rilzabrutinib
Description: Plasma samples were collected at specified timepoints to determine CL/F of rilzabrutinib.
Time Frame: Day 1 of Cycles 1, 2, and 3 (each cycle 28 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | Part A: Dose Level 200 mg QD | Part A: Dose Level 400 mg QD | Part A: Dose Level 300 mg BID | Part A: Dose Level 400 mg BID
Number analyzed (Participants) | 9 | 5 | 7 | 35
liters/hour
  Cycle 1 Day 1: number analyzed (Participants) | 9 | 0 | 5 | 35
  Cycle 1 Day 1 | 911 (569) |  | 592 (320) | 854 (551)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 5 | 0 | 1
  Cycle 2 Day 1 |  | 743 (593) |  | 484 (NA) — SD cannot be calculated for a single participant.
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 7 | 0
  Cycle 3 Day 1 |  |  | 713 (621) |

26. Secondary Outcome: Part B: Plasma Concentration of Rilzabrutinib
Description: Plasma samples were collected at specified timepoints for evaluation of rilzabrutinib pharmacokinetic (PK) concentrations.
Time Frame: Pre-dose and 2 hours post-dose on Days 1, 29, and 57
Population: PK population consisted of all enrolled participants from the safety population who had at least 1 post-baseline PK result.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B: Rilzabrutinib 400 mg BID
Number analyzed (Participants) | 25
ng/mL
  Day 1: pre-dose | NA (NA) — Mean and SD were not calculated as the values were below the lower limit of quantification (LLOQ=0.100 ng/mL).
  Day 1: 2 hours post-dose | 154.09 (131.79)
  Day 29: pre-dose: number analyzed (Participants) | 22
  Day 29: pre-dose | 5.07 (8.61)
  Day 29: 2 hours post-dose: number analyzed (Participants) | 23
  Day 29: 2 hours post-dose | 228.67 (173.68)
  Day 57: pre-dose: number analyzed (Participants) | 22
  Day 57: pre-dose | 26.42 (90.43)
  Day 57: 2 hours post-dose: number analyzed (Participants) | 22
  Day 57: 2 hours post-dose | 331.81 (151.07)

ADVERSE EVENTS:
Time Frame: Adverse events data was collected from first dose of rilzabrutinib (Day 1) up to last dose + 1, approximately up to 294 days (Part A) and up to 170 days (Part B). All-cause mortality (death) was assessed from the signing of the ICF up to primary completion date (31 January 2023) approximately 253 weeks.
Description: Analysis was performed on safety population. As pre-specified (SAP), AEs were presented by dose level and overall . A participants could be classified into multiple dose levels.
Groups:
- Part B: 400 mg BID: Participants received rilzabrutinib 400 mg orally BID from Day 1 up to 24 weeks of treatment period.
Arm/Group | Part A: Dose Level 200 mg QD | Part A: Dose Level 400 mg QD | Part A: Dose Level 300 mg BID | Part A: Dose Level 400 mg BID | Part A: Overall | Part B: 400 mg BID
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/12 | 1/52 | 1/60 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/8 | 3/12 | 9/52 | 11/60 | 3/26
Other Adverse Events (participants affected / at risk) | 5/9 | 6/8 | 9/12 | 43/52 | 48/60 | 21/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Dose Level 200 mg QD (N=9) | Part A: Dose Level 400 mg QD (N=8) | Part A: Dose Level 300 mg BID (N=12) | Part A: Dose Level 400 mg BID (N=52) | Part A: Overall (N=60) | Part B: 400 mg BID (N=26)
Covid-19 Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Evans Syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Immune Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Dose Level 200 mg QD (N=9) | Part A: Dose Level 400 mg QD (N=8) | Part A: Dose Level 300 mg BID (N=12) | Part A: Dose Level 400 mg BID (N=52) | Part A: Overall (N=60) | Part B: 400 mg BID (N=26)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (6)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 5 (6) | 4 (5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 4 (6) | 2 (3)
Haemorrhagic Diathesis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abnormal Dreams (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 7 (9) | 7 (9) | 9 (13)
Conjunctival Haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 5 (6) | 5 (6) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ear Pruritus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 4 (5)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 6 (6) | 6 (6) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 5 (6)
Aphthous Ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 22 (30) | 23 (31) | 12 (16)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 4 (5) | 5 (6)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Gingival Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 3 (5) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Loose Tooth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 19 (25) | 21 (27) | 7 (11)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (5) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 2 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 4 (5) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 6 (9) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 9 (11) | 10 (12) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Micturition Urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 2 (2) | 12 (14) | 13 (15) | 3 (3)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Peripheral Swelling (General disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
Vessel Puncture Site Bruise (General disorders) | 1 (2) | 1 (2) | 1 (2) | 1 (2) | 1 (2) | 0 (0)
Vessel Puncture Site Discharge (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 3 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (7) | 3 (7) | 3 (7) | 10 (18) | 12 (20) | 5 (10)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT03395210/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT03395210/SAP_001.pdf